CLINICAL TRIAL: NCT01682642
Title: IVF Outcome in Patients With Peritoneal Endometriosis. The Impact of a Hormonal Treatment of the Endometriosis Prior to the IVF on the Pregnancy Rates.
Brief Title: The Influence of Adjuvant Medical Treatment of Peritoneal Endometriosis on the Outcome of IVF. A Prospective Randomized Analysis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AZ Jan Palfijn Gent (Other)
Collaborators: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Dr. Decleer Wim, gynecologist, AZ Jan Palfijn Gent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-000784-25
Record Dates: First submitted 2012-08-23; First posted 2012-09-11 (Estimated); Results first posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Infertility; Endometriosis
Keywords: endometriosis; pregnancy; In Vitro Fertilization (IVF)/Intra Cytoplastic Sperm Injection (ICSI); peritoneal implants; embryo quality
MeSH Terms: conditions — Infertility; Endometriosis | interventions — Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoladex (Active Comparator): After surgical vaporization of endometriosis patients are treated with Zoladex for 3 months.
  Interventions: Drug: Zoladex
- vaporization only (No Intervention): Surgical vaporization of the endometriosis is done and patients start IVF without additional treatment.

INTERVENTIONS:
Drug: Zoladex — after surgical vaporization patients are treated with Zoladex for 3 months before starting IVF treatment
  Arms: Zoladex

SUMMARY:
In this study of endometriosis patients we compare a common treatment of surgical therapy and medical treatment for 3 months (Zoladex) with patients receiving only surgical therapy. In both cases they immediately start In Vitro Fertilization (IVF) treatment.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopical vaporization of endometriosis
* 1,2, 3e IVF cycle
* endometriosis stage I and II
* younger than 38 years

Exclusion Criteria:

* endometriosis cysts
* uterine pathology
* endocrinological diseases and problems

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wim Decleer, gynecologist, Principal Investigator — Fertility Center AZ Jan Palfijn Gent; Paul Devroey, Professor, Study Chair — Fertility Center AZ Jan Palfijn Gent
Locations (1):
- AZ Jan Palfijn, Ghent, Oost-vlaanderen, Belgium

RESULTS

PARTICIPANT FLOW:
Groups:
- Zoladex: After surgical vaporization of endometriosis, patients are treated with Zoladex for 3 months immediately following the start of IVF treatment.
- Vaporization Only: After surgical vaporization of the endometriosis , patients start immediately with IVF treatment (without additional treatment).
Period: Overall Study
Arm/Group | Zoladex | Vaporization Only
Started | 61 | 59
Completed | 61 | 58
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: women between 18 and 38 years
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoladex | Vaporization Only | Total
Number analyzed (Participants) | 61 | 58 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 58 | 119
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.33 (3.63) | 31.70 (4.28) | 31.02 (3.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 58 | 119
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 61 | 58 | 119

OUTCOME MEASURES:

1. Primary Outcome: Number of Metaphase II Cells (MII)
Description: number of MII cells retrieved
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: MII cells
Arm/Group | Zoladex | Vaporization Only
Number analyzed (Participants) | 61 | 58
MII cells | 8.2 (5.92) | 8.2 (4.82)

2. Secondary Outcome: Pregnancy Rate
Description: The number of ongoing pregnancies obtained which still is the most important issue for the patients.
Time Frame: 12 weeks
Measure: Number; unit: percentage of ongoing pregnancies
Arm/Group | Zoladex | Vaporization Only
Number analyzed (Participants) | 61 | 58
percentage of ongoing pregnancies | 39.3 | 39.7

3. Secondary Outcome: Good Embryo Quality
Description: The development of the embryo at the time of transfer on day 3. Good quality is defined by more than 7 cells and less then 20% fragmentation on day 3.
Time Frame: 3 days after oocyte retrieval
Measure: Number; unit: percentage of good quality embryos
Groups:
- Zoladex: After surgical vaporization of endometriosis, patients are treated with Zoladex for 3 months and immediately following start of IVF treatment.
Arm/Group | Zoladex | Vaporization Only
Number analyzed (Participants) | 61 | 58
percentage of good quality embryos | 59.3 | 67.3

4. Secondary Outcome: Number of Pro Nuclear Cell (2PN)
Description: number of 2PN
Time Frame: 1 day after oocyte retrieval
Measure: Mean (Standard Deviation); unit: number of pro nuclear cells
Arm/Group | Zoladex | Vaporization Only
Number analyzed (Participants) | 61 | 58
number of pro nuclear cells | 5.4 (4.03) | 5.6 (4.20)

5. Secondary Outcome: Number of Cryopreserved Embryos
Description: number of blastocytes that can be cryopreserved
Time Frame: 1 week after oocyte retrieval
Measure: Mean (Standard Deviation); unit: number of cryopreserved embryos
Groups:
- Zoladex: After surgical vaporization of endometriosis, patients are treated with Zoladex for 3 months and immediately following start of IVFtreatment.
- Vaporization Only: Surgical vaporization of the endometriosis is done and patients immediately start IVF without additional treatment.
Arm/Group | Zoladex | Vaporization Only
Number analyzed (Participants) | 61 | 58
number of cryopreserved embryos | 0.9 (1.40) | 1.6 (2.31)

6. Other Pre Specified Outcome: Number of Days of Stimulation
Description: number of days needed before follicles in the ovary are mature for oocyte retrieval
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: days
Groups:
- Zoladex: After surgical vaporization of endometriosis, patients are treated with Zoladex for 3 months and immediately following start IVF treatment.
Arm/Group | Zoladex | Vaporization Only
Number analyzed (Participants) | 61 | 58
days | 12.3 (1.86) | 11.3 (1.98)

7. Secondary Outcome: Total Follicle Stimulating Hormone (FSH) Dose
Description: total dose of FSH needed at the end of stimulation
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: IUs
Groups:
- Zoladex: After surgical vaporization of endometriosis, patients are treated with Zoladex for 3 months and immediately following ivf treatment.
Arm/Group | Zoladex | Vaporization Only
Number analyzed (Participants) | 61 | 58
IUs | 2561 (621.7) | 2303 (604.8)

ADVERSE EVENTS:
Arm/Group | Zoladex | Vaporization Only
Serious Adverse Events (participants affected / at risk) | 11/61 | 7/58
Other Adverse Events (participants affected / at risk) | 1/61 | 0/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoladex (N=61) | Vaporization Only (N=58)
OHSS (Reproductive system and breast disorders) | 11 | 7 — Ovary Hyper Stimulation Syndrome (OHSS)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoladex (N=61) | Vaporization Only (N=58)
miscarriage (Surgical and medical procedures) | 1 (1) | 0 (0) — pregnancy lost in first trimester

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No